CLINICAL TRIAL: NCT05656508
Title: Phase 1 Study to Evaluate Safety, Tolerability and Immunogenicity of a New Recombinant Protein-based Vaccine (ARVAC CG) Against Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2), in a Population of Healthy Adult Volunteers Previously Vaccinated Against SARS-CoV-2 Virus.
Brief Title: ARVAC - A New Recombinant Coronavirus Disease 2019 (COVID-19) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorio Pablo Cassara S.R.L. (Industry)
Collaborators: Universidad Nacional de San Martín (UNSAM) (Unknown); National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARVAC-F1-001
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Vaccine

STUDY DESIGN:
Intervention Model Description: The volunteers will be divided into 2 arms:
  Group 1 will receive a vaccination schedule of 2 doses of 25 µg of antigen Group 2 will receive a vaccination schedule of 2 doses of 50 µg of antigen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 µg of antigen (Experimental): Volunteers will receive 2 doses of ARVAC-CG vaccine (recombinant protein vaccine against SARS-CoV-2) of 25 µg of antigen, separated by 28 days
  Interventions: Biological: ARVAC-CG vaccine (recombinant protein vaccine against SARS-CoV-2)
- 50 µg of antigen (Experimental): Volunteers will receive 2 doses of ARVAC-CG vaccine (recombinant protein vaccine against SARS-CoV-2) of 50 µg of antigen, separated by 28 days
  Interventions: Biological: ARVAC-CG vaccine (recombinant protein vaccine against SARS-CoV-2)

INTERVENTIONS:
Biological: ARVAC-CG vaccine (recombinant protein vaccine against SARS-CoV-2) — 2 doses of vaccine with an interval between doses of 28 days. Administration route: Intramuscular (IM) injection

SUMMARY:
The objective of this clinical trial is to test a new vaccine against SARS-CoV-2 (ARVAC-CG) in healthy adult volunteers, previously vaccinated against the SARS-CoV-2 virus.

The main questions it aims to answer are:

* What is the safety and tolerability profile of the two-dose schedule of this new vaccine?
* What is the immune response after each dose of vaccine Participants will receive two doses of the study vaccine 28 days apart. They will be required to complete a total of 7 safety and immunogenicity follow-up visits over a 1-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 55 years of age
2. With the ability and willingness to comply with the prohibitions and restrictions specified in the protocol.
3. Healthy volunteers, which will be determined by the history referred to interrogation, physical examination, and principal investigator's criteria.
4. In fertile female volunteers, negative pregnancy test at the beginning of the study and commitment to use a contraceptive method from the date of signing the consent form until 3 months after vaccine study application. Use of a hormonal contraceptive method must begin at least 28 days prior to study vaccine application. The investigator should assess potential contraceptive method failure (e.g. non-compliance, recent onset) in relation to vaccination. Acceptable effective methods for this study include:

   a) hormonal contraceptive method: i) combined (containing estrogen and progestin) associated with the inhibition of ovulation (oral, intravaginal or transdermal); ii) with progestin only, associated with the inhibition of ovulation (oral, injectable or implantable); b) intrauterine device;. c) intrauterine hormone release system; d) bilateral tubal ligation/occlusion procedure; e) single couple with vasectomy; f) sexual abstinence, which will be considered effective only if it is defined as abstaining from heterosexual relations from the date of signing the consent until 3 months after receiving the study vaccine. The reliability of sexual abstinence should be assessed in relation to the duration of the study and the participant's usual and preferred lifestyle.
5. Participant who agrees to do not donate bone marrow, blood or blood products until 3 months after the last dose of study vaccine;
6. Participant who is able to read, understand, and complete electronic questionnaires about signs and symptoms of COVID-19 surveillance;
7. Negative PCR for the SARS-CoV-2 virus.
8. With laboratory analysis without clinically significant variations within the 30 days prior to receiving the first dose of the study vaccine, which must include:

   1. complete cell blood count (hemoglobin (Hb), leukocyte count and leukocyte formula, platelet count;
   2. complete liver test: total and direct bilirubin, alanine aminotransaminases (ALT) and aspartate aminotransferase (AST), lactate dehydrogenase (LDH), alkaline phosphatase (ALF).
   3. biochemistry: glycemia, urea, creatinine;
   4. Qualitative C-reactive protein (PCR);
   5. Complete urine.
9. Capable of granting their informed consent signed and dated by the volunteer under study, and the authorized physician.

Exclusion Criteria:

1. History of SARS-CoV-2 infection or known previous disease, within 60 days prior to study entry (at least 60 days from epidemiological discharge).
2. Administration of any other commercial vaccine or not, based on:

   1. Live attenuated virus within 28 days prior to study entry.
   2. Killed virus within 14 days prior to study entry.
3. Individuals that have not received a complete primary vaccination schedule against SARS-CoV-2 virus (1 or 2 doses, depending on the vaccine used in the primary schedule).
4. Administration of complete primary vaccination schedule against SARS-CoV-2 virus (1 or 2 doses, depending on the vaccine received), within 4 months prior to the start of the study.
5. Administration of an additional or booster dose after a complete primary vaccination schedule against SARS-CoV-2 virus.
6. Individuals that have scheduled to receive any other commercial vaccine in the following 3 months.
7. Individuals that have participated in a research study within 60 days prior to the start of the study.
8. History of known allergies or a history of anaphylaxis or any other serious adverse reaction with other vaccines or their excipients.
9. History of alcoholism or substance abuse that prevents compliance with the characteristics of the protocol.
10. Acute infectious disease at enrollment (this does not include minor conditions such as diarrhea or mild upper respiratory tract illness) or temperature ≥38. 0°C within 24 hours prior to scheduled study vaccination; later admission is permitted at the discretion of the investigator and after the Sponsor agreement.
11. Any laboratory determination alteration with a degree of severity > 1 according to the Common Toxicity Criteria (CTC version 5 - November 2017). Participants with any stable grade 1 abnormality may be considered eligible by the investigator. (grade 1 stable implies a repetition of the sample that persists with an alteration of one grade no greater than 1).
12. Body Mass Index (BMI) greater than 30 kg/m2 or less than 18 kg/m2.
13. Individuals currently working in occupations with high exposure to SARS-CoV-2.
14. History of any clinical condition that affects the function of the immune system, including, but not limited to:

    1. Clinical conditions (e.g. autoimmune disease or possibly immune-mediated disease or known or suspected immunodeficiency; diabetes mellitus type I or II, chronic kidney disease, etc.).
    2. Chronic or recurrent use of systemic corticosteroids in the 6 months prior to study vaccine administration and during the study. A substantially immunosuppressive dose of steroids is considered ≥2 weeks of daily administration of 20 mg prednisone or equivalent.
    3. Administration of antineoplastic and immunomodulatory agents or radiation therapy within 6 months prior to study vaccine administration or during the study.
15. The volunteer has received an investigational drug (including drugs related to COVID-19 prophylaxis) or used an investigational invasive medical device in the past 30 days or has received investigational immunoglobulin or monoclonal antibodies within 3 months (participation in an observational study is allowed at the discretion of the investigator, previously informing the Sponsor about this decision).
16. The participant is pregnant, plans to become pregnant within 3 months after the administration of the vaccine, or is in postpartum or lactation period.
17. The volunteer has any contraindication to receive intramuscular injections and/or blood draws.
18. The volunteer has a history of acute polyneuropathy (e.g. Guillain Barré syndrome).
19. The volunteer underwent a surgical procedure that required hospitalization (defined as hospitalization for more than 24 hours or overnight hospitalization), in the 12 weeks prior to vaccination, or has not recovered completely from surgery that required hospitalization or is scheduled for surgery that will require hospitalization during the time he/she is expected to participate in the study or within 6 months of study vaccine administration.
20. Positive serology for hepatitis (Hepatitis B surface antigen [HBsAg], Hepatitis B core antigen antibodies [Anti-HBc], Hepatitis C virus antibodies [Anti-HCV]).
21. Positive antibodies against Human Immunodeficiency Virus (HIV).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Safety: Solicited local and systemic reactions after administration of each dose of the vaccine. | Day 0 to 7 after each vaccination
  Number of volunteers overall and in each dose group with local or systemic vaccine reactogenicity, based on evaluation of solicited adverse events (AEs) recorded on subject memory aids or during clinical assessments
Safety: Unsolicited adverse events after each vaccine dose | Day 0 to 30 after each vaccination
  Number of volunteers overall and in each dose group with unsolicited vaccine-associated adverse events (AEs) in each dose group
Safety: Serious adverse events | Day 0 to 30 after each vaccination
  Number of volunteers overall and in each dose group with vaccine-associated serious adverse events (SAEs)
Safety: Variations in the laboratory results | Day 0 to 56 after vaccination
  Number of volunteers overall and in each dose group with variations in laboratory results from a baseline control at days 7, 28 and 56.

SECONDARY OUTCOMES:
Immunogenicity: Neutralizing antibodies | Day 0 to 28 days after each vaccine dose
  Geometric Mean Title (GMT) at baseline, 14 days and 28 days after each dose
Immunogenicity: Total specific antibodies | Day 0 to 28 days after each vaccine dose
  Geometric Mean Title (GMT) at baseline and 28 days after each dose
Immunogenicity: Number of Inteferon (IFN) gamma and interleukin (IL)-4 producing cells directed to Receptor Binding Domain (RBD) (Spike protein region) | Day 0 to 28 days after each vaccine dose
  Determination of cellular immune response, specific IFN gamma and IL-4 producing cells directed to RBD (Spike protein region) on day 1 (prior to the first dose) and 28 days after each vaccine dose

OTHER OUTCOMES:
Exploratory variables: Neutralizing antibodies titer variation according to primary vaccination schedule | Day 0 to 28 days after each vaccine dose
  Variation of GMT of neutralizing antibodies between day 0, day 14 and day 28 after each dose, according to the primary vaccination schedule received
Exploratory variables: Neutralizing antibodies titer variation according to vaccine platform used in the primary scheme | Day 0 to 28 days after each vaccine dose
  Variation of GMT of neutralizing antibodies between day 0, day 14 and day 28 after each dose, depending on vaccine platform used in the primary scheme
Exploratory variables: Neutralizing antibodies titer variation according to dose of the study vaccine received | Day 0 to 28 days after each vaccine dose
  Variation of GMT of neutralizing antibodies between day 0, day 14 and day 28 after each dose, depending on the dose of the study vaccine received (2 doses of 25 µg of antigen or 2 doses of 50 µg of antigen).
Exploratory variables: Neutralizing antibodies titer variation according to history of having had a previous SARS-CoV-2 infection or not | Day 0 to 28 days after each vaccine dose
  Variation of GMT of neutralizing antibodies between day 0, day 14 and day 28 after each dose, depending on history of having had a previous SARS-CoV-2 infection or not

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A YERINO, MD., Principal Investigator — Unidad de Investigación Clínica Farmacocinética FP Clinical Pharma en Clínica CIAREC
Locations (1):
- Unidad de Investigación Clínica Farmacocinética FP Clinical Pharma en Clínica CIAREC, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: all of the individual participant data collected during the trial after deidentification and after publication of the results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available immediately following publication
Access Criteria: Access will be given to researchers who provide a methodologically sound proposal or whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Proposals should be directed to the corresponding author of the publication.

REFERENCES:
- [Derived] Pasquevich KA, Coria LM, Ceballos A, Mazzitelli B, Rodriguez JM, Demaria A, Pueblas Castro C, Bruno L, Saposnik L, Salvatori M, Varese A, Gonzalez S, Gonzalez Martinez VV, Geffner J, Alvarez D; Laboratorio Pablo Cassara R&D and CMC for ARVAC CG consortium; Feleder E, Halabe K, Perez Lera PE, de Oca FM, Vega JC, Lombardo M, Yerino GA, Flo J, Cassataro J. Safety and immunogenicity of a SARS-CoV-2 Gamma variant RBD-based protein adjuvanted vaccine used as booster in healthy adults. Nat Commun. 2023 Jul 28;14(1):4551. doi: 10.1038/s41467-023-40272-3. PMID 37507392